CLINICAL TRIAL: NCT01160978
Title: Donor Simvastatin Treatment in Organ Transplantation
Acronym: SIMVA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Academy of Finland (Other)
Responsible Party: Principal Investigator, Karl Lemstrom, Consultant Cardiothoracic Surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T1020SIMVASTATIN
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure; Respiratory Failure; Liver Failure; Kidney Failure; Transplantation
Keywords: Transplantation; Simvastatin treatment; Ischemia-reperfusion injury; Rejection
MeSH Terms: conditions — Heart Failure; Respiratory Insufficiency; Liver Failure; Renal Insufficiency; Reperfusion Injury; Rejection, Psychology | interventions — Simvastatin; Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin 80 mg group (Active Comparator): The transplant recipients who have received an organ from donors treated with simvastatin 80 mg.
  Interventions: Drug: Simvastatin 80mg
- Control Rx (Experimental): The transplant recipients who have received an organ from non-treated donors.
  Interventions: Drug: Control Rx

INTERVENTIONS:
Drug: Simvastatin 80mg — The transplant recipients who have received an organ from donors treated with simvastatin 80 mg.
  Other Names: simvastatin
  Arms: Simvastatin 80 mg group
Drug: Control Rx — The transplant recipients who have received an organ from non-treated donors.
  Arms: Control Rx

SUMMARY:
The aim of the study is to investigate the effects of donor simvastatin treatment on ischemia-reperfusion injury after heart transplantation.

DETAILED DESCRIPTION:
The study hypothesis of the single center randomized double-blinded clinical trial is that donor simvastatin treatment reduces ischemia-reperfusion injury after heart transplantation. Also, it potentially decreases natural immune activity, rejection activation and thus improves long-term prognosis.

Simvastatin is administered to heart and/or lung donors through the nasogastric tube 4-6 hours prior to organ harvesting. Control organ donors do not receive simvastatin. The randomization and donor hospital instruction of the donor simvastatin treatment is performed by the transplant coordinator. All other caregivers and the transplant recipient are blinded to the treatment group allocation.

The impact of donor simvastatin treatment is investigated and analyzed by several specific blood samples and biopsies that are taken from the recipient at the various time-points during the perioperative and postoperative phase.

In heart transplant recipients (n=42 in the donor simvastatin treatment group and n=42 in the control group), the primary end-point is postoperative cardiac enzyme serum levels (TnT, TnI, and CK-MB 1 hour, 6 hours, 12 hours and 24 hours after transplantation) and primary graft failure. Secondary end-points include peri- and postoperative parameters hemodynamics, short- and long term survival, biopsy-proven rejections, rejection treatments, and chronic rejection at 1, 5, 10, and 20 years after transplantation.

Lung, kidney and liver transplant recipients that have received organs from donors randomized to the control group or donor simvastatin group will also be followed for ischemia-reperfusion injury, perioperative organ function, innate and adaptive immunity and patient survival.

ELIGIBILITY:
Inclusion criteria for a donor:

* Heart transplant donor
* Age 18-60 years
* Previously healthy
* No cholesterol medication
* Normal ECHO with LVEF >45%, normal right ventricle and normal coronary angiography
* PiO2/FiO2 > 40kPA, normal chest radiograph and normal bronchoscopy in lung donors

Exclusion Criteria for the heart/lung donor:

* Severe left ventricular hypertrophy > 14 mm
* High dose of inotropes (dopamine or dobutamine > 20ug/kg/min or norepinephrine >0.2 ug/kg/min) at the time of procurement
* Donor outside of the study country Finland

Inclusion criteria for a transplant recipient:

* Age between 18-70 for heart transplant recipients
* Male or female
* Listed for heart, lung, kidney, or liver transplantation

Exclusive Criteria for the recipient

* systemic sepsis
* a positive cross match

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Donor treatment with simvastatin reduces ischemia-reperfusion injury after heart transplantation | 1-24 hour
  Recipient plasma release of cardiac troponins and creatinine kinase-MB and P-lactate, S-hs-CRP, peripheral blood leukocytes and neutrophils after heart transplantation

SECONDARY OUTCOMES:
Postoperative hemodynamics | 0-72h
  Arterial line and pulmonary artery catheter measurements 6, 12, 24, 48, and 72 hours
Postoperative use of inotropes and hemodynamic support | 0-72h
  Postoperative use of inotropes and hemodynamic support at 6, 12, 24, 48, and 72 hours and the length of inotropic support
Heart transplant function | 0-20 years
  Heart transplant function analyzed by P-ProBNP and echocardiogram
Cardiac allograft vasculopathy | at 1, 3, and 5 years
  Cardiac allograft vasculopathy analyzed coronary angiogram
Biopsy proven acute rejection | 0-20 years
  Grade of rejection at endomyocardial biopsy
Rejection treatments | 0-20 years
  Any rejection treatments
Short- and long-term survival | 0-20 years
  Time to all-cause mortality
Substudy 1 | 0-20 years
  Outcome of kidney transplant recipients
Substudy 2 | 0-20 years
  Outcome of liver transplant recipients
Substudy 3 | 0-20 years
  Outcome of lung transplant recipients
Substudy 4 | 0-24 h
  Development of biomarkers for ischemia-reperfusion injury after heart transplantation
Substudy 5 | 0-1 years
  Development of molecular profiling for endomyocardial biopsy after heart transplantation
Substudy 6 | 0-20 years
  Effect of donor and recipient genomic backgroud on long term outcomes after heart transplantation
Substudy 7 | 0-20 years
  Effect of donor and recipient genomic backgroud on long term outcomes after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Karl B Lemstrom, MD, PhD, Principal Investigator — Cardiac surgery, Heart and Lung Center, Helsinki University Hospital
Locations (1):
- Cardiac Surgery, Heart and Lung Center, Helsinki University Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Nykanen AI, Holmstrom EJ, Tuuminen R, Krebs R, Dhaygude K, Kankainen M, Jokinen JJ, Lommi J, Helantera I, Raisanen-Sokolowski A, Syrjala SO, Lemstrom KB. Donor Simvastatin Treatment in Heart Transplantation. Circulation. 2019 Aug 20;140(8):627-640. doi: 10.1161/CIRCULATIONAHA.119.039932. Epub 2019 Jul 29. PMID 31352795
- See also: Website of Heart and Lung Center, Helsinki University Hospital — http://www.hus.fi/sydanjakeuhkokeskus
- See also: Website of Transplantation Laboratory, University of Helsinki — https://www.helsinki.fi/en/researchgroups/transplantation-laboratory